CLINICAL TRIAL: NCT04852393
Title: A Prospective Evaluation of the Safety and Clinical Effects of Ultrasound-guided Cervical Medial Branch Blocks
Brief Title: Ultrasound-guided Cervical Medial Branch Blocks
Status: Completed | Type: Observational
Sponsor: Montreal General Hospital (Other)
Responsible Party: Principal Investigator, Roderick Finlayson, Professor, University of British Columbia
Other Study IDs: 2020-21-105-H
Record Dates: First submitted 2021-04-12; First posted 2021-04-21 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Neck Pain; Cervical Spondylosis
MeSH Terms: conditions — Neck Pain; Spondylosis | interventions — Dental Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Block: Patients undergoing ultrasound-guided cervical medial branch blocks as part of their usual care
  Interventions: Procedure: Block

INTERVENTIONS:
Procedure: Block — cervical medial branch block

SUMMARY:
In this study we will prospectively examine the safety and clinical effects of ultrasound-guided cervical medial branch blocks.

DETAILED DESCRIPTION:
While several clinical trials have found that ultrasound guidance provides similar accuracy to fluoroscopy and reduces performance times for cervical medial branch blocks, larger studies documenting safety-related outcomes are lacking. In addition, although cervical medial branch blocks are an accepted tool to diagnose neck pain originating from the cervical facets, there are reports of long-lasting analgesic effects in a subset of patients, suggesting that these blocks may have long-term benefits. We therefore propose to prospectively examine the incidence of adverse events, as well as the clinical long-term effects of ultrasound-guided cervical medial branch blocks, in a cohort of pain clinic patients undergoing these procedures as part of their usual care.

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients over 18 years of age undergoing cervical medial branch blocks as part of their usual care and who have a pain intensity of at least 5/10 (at rest or on movement) and a pain duration of at least 4 months.

Exclusion Criteria:

* Inability to communicate or complete follow up questionnaires
* Known bleeding disorder or coagulopathy
* Patients on antiplatelet medication other than aspirin and those on anticoagulants (coumadin, AT III agents)
* Inability to visualize targeted structures on ultrasound
* Presence of acute radiculopathy of new onset neurological symptoms in the upper extremities
* Patients with bilateral neck pain if only one side is treated

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to a tertiary outpatient pain clinic for diagnosis and treatment of chronic neck pain
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Immediate complications | Immediately after block
  Proportion of patients with immediate block-related complications including any of the following: vasovagal, local anesthetic toxicity (dizziness, tinnitus, altered LOC, seizure) and trauma to non-targeted neural structures (paresthesia or other neuro symptoms)
Delayed complications | 14 days after block
  Proportion of patients with delayed block-related complications including any of the following: redness/irritation/swelling at injection site, hematoma, infection, skin bruising, soreness at injection site or increased pain, any neurological symptoms (new onset radicular pain, numbness/weakness or paresthesia in upper extremities).

SECONDARY OUTCOMES:
Patient reported pain | Pre-block, then every 2 weeks for 3 months.
  Lowest/highest/average pain score over last 7 days (NRS, 11-point scale)
NDI | Pre-block, then every 2 weeks for 3 months.
  Neck disability index
PHQ-9 | Pre-block then at 1,2 and 3 months post block.
  Depression scale
GAD-7 | Pre-block then at 1,2 and 3 months post block.
  Anxiety scale
PCS | Pre-block then at 1,2 and 3 months post block.
  Pain catastrophizing scale
PGIC | Pre-block, then every 2 weeks for 3 months.
  Patient global impression of change 7-point scale

CONTACTS AND LOCATIONS:
Overall Officials: Roderick J Finlayson, MD, Principal Investigator — University of British Columbia; John-Paul B Etheridge, MD, Principal Investigator — University of British Columbia
Locations (1):
- Bill Nelems Pain and Research Centre, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Finlayson RJ, Etheridge JB, Godard R, Kaseweter K, Etheridge JP, Curatolo M. Do cervical medial branch blocks have a therapeutic role? a prospective cohort study. Reg Anesth Pain Med. 2025 May 28:rapm-2025-106457. doi: 10.1136/rapm-2025-106457. Online ahead of print. PMID 40441772
- [Derived] Etheridge JB, Finlayson RJ, Venter J, De Villiers F, Etheridge JP, Wakefield R, Watanitanon A. Prospective evaluation of the safety of ultrasound-guided cervical medial branch blocks using the in-plane technique. Reg Anesth Pain Med. 2025 Mar 5;50(3):237-242. doi: 10.1136/rapm-2024-105296. PMID 38508589